CLINICAL TRIAL: NCT00853775
Title: Regulation of Lipoprotein(a) Metabolism in Humans With Reference to Ethnicity
Brief Title: Family Research Study: Metabolism of Fats and Proteins in Specific Ethnic Groups
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 200816533; 2R01HL062705-05A2 (NIH)
Record Dates: First submitted 2009-02-25; First posted 2009-03-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Heart Disease
Keywords: heart disease; cardiovascular disease; lipoproteins; lipoprotein(a); Lp(a); apolipoprotein(a); apo(a); fats; proteins; metabolism
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma, DNA, white blood cell
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- African American Families: Families with 2 parents and 2 children - no intervention, observational study
  Interventions: Other: No intervention, observational study
- Caucasian Families: Families with 2 parents and 2 children - no intervention, observational study
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study

SUMMARY:
The purpose of this study is to determine whether lipoprotein(a), also called Lp(a), is a risk factor for cardiovascular (heart) disease. Lipoproteins are tiny particles that circulate in the blood. They contain cholesterol, fat, and protein in varying amounts depending on the body's need. Higher levels of lipoproteins in the blood can cause an increased risk of heart disease.

The investigators believe that by studying the Lp(a) lipoprotein in Caucasians and African Americans, the investigators can assess for genetic variation factors related to cardiovascular (heart) disease. The investigators will be looking at 100 African-American families and 100 Caucasian families to confirm whether a higher Lp(a) level is an indicator of a higher risk for heart disease.

DETAILED DESCRIPTION:
During the study visit the research staff will ask about the medical history, perform a brief physical exam, and draw approximately 4 teaspoons of blood of each family member.

ELIGIBILITY:
Inclusion Criteria:

* Of Caucasian or African descent
* Families must have 2 natural/biological parents and 2 natural/biological offspring
* 6 years old or older

Exclusion Criteria:

* Races other than African American or Caucasian
* Families without 2 natural/biological parents and 2 natural/biological offspring
* younger that 6 years old

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We are recruiting 100 African American and 100 Caucasian families. The families that will be recruited will have two natural parents and two natural offspring.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Genetic variation of Lp(a) levels in each group | five years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Berglund, M.D., Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis CTSC Clinical Research Center (CCRC) at Veterans Affair Medical Center, Mather, California, United States